CLINICAL TRIAL: NCT02255708
Title: Electromyography Evaluation of the Stabilizing Muscles of the Scapula and Tibial Anterior Muscle, After an Intervention Program by Proprioceptive Neuromuscular Facilitation in Muscle Force Irradiation.
Brief Title: Effects of an Intervention Program by Proprioceptive Neuromuscular Facilitation, in Muscle Force Irradiation.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Cláudia Silva Ferreira, Ana Cláudia Silva Ferreira, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1161-5560
Record Dates: First submitted 2014-09-23; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Assessment of Muscle Force Irradiation
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy group. (Other): Group formed by healthy patients.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation - PNF
- Group with demyelinating polyneuropathy (Other): Group formed by patients with demyelinating polyneuropathy.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation - PNF

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation - PNF

SUMMARY:
The present study aims to assess through surface electromyography, the effectiveness of proprioceptive neuromuscular facilitation protocols in the activation of the stabilizing muscles of the scapula and the anterior tibial muscle.

DETAILED DESCRIPTION:
Healthy subjects and subjects with demyelinating polyneuropathy are involved in the study.

Healthy patients are arranged in two groups of stimulation: FNP Group (intervention proprioceptive neuromuscular facilitation) - CC Group (intervention classic cinesioterapia). The electromyographic response of the stabilizing muscles of the scapula of each individual will be assessed prior to application of the protocols, during the execution of the protocols and immediately after stopping in a single session.

Patients with demyelinating polyneuropathy are arranged in a single treatment group and will be treated at a frequency of twice a week for five weeks. In each session, the PNF patterns will be repeated four times, on both sides, stimulating muscle irradiation and evoking the contraction of the tibialis anterior muscle. During the repetition of the patterns, the dorsiflexor muscle response of each patient will be obtained by an electromyography (EMG) surface.

The data of the RMS values obtained in the first session will be normalized and transformed into percentage. The average RMS of each diagonal at the beginning of treatment corresponds to 100% of TA muscle activation. The RMS values obtained in the last session will be normalized as a percentage, taking into account the results of the first evaluation. After normalization, data from the first and last sessions will besubjected to the for paired t-test.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals group: who agree to participate in the study with no history of previous trauma or disease of the shoulder girdle, with absence of clinical signs painful in the shoulder joint.

Group with demyelinating polyneuropathy: both sexes, carriers of CMT-1A disease with functional changes in the lower limbs with good cognition and difficulty of to ambulate with and without assistance.

Exclusion Criteria:

Healthy individuals group: subject with restricted range of motion, muscle weakness, cognitive impairment, which exhibits a pathology that leads to alterations in muscle recruitment.

Patients with polyneuropathy: cardiac arrhythmias, uncontrolled hypertension, severe cardiovascular disease and respiratory problems. The use of own medicines to treat pathology was accepted.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of muscle force irradiation, through surface electromyography. | This evaluation of patients is performed in only one day, being made before, during and after the application of the protocols. It is estimated that the results are collected in one years.
  Irradiation of muscle strength will be assessed using surface electromyography, which shows the activation or not of the muscles evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Neuropsychobiology and Motor Behavior,, Ribeirão Preto, São Paulo, Brazil